### Balanced Nutritional Diet Intervention on Body Composition Among Different FTO RS9939609 Gene in Obese Young Women In Bandung, Indonesia: A Randomised Controlled Trial

Update 10 October 2023

No. Register: 7 0 3 6 1 0 8 9 **General information** A. Putri Novitasari, S.Gz., M.Si 1. Principal Researcher (Name and title) Skills/Specialization **Nutrition Science** Position/Position IPB Doctoral Student (S3) e-mail: putrinovitasarigizi@gmail.com Tel. House: -MOBILE PHONE: 08112227291 2. Origin of Institution: Non-Unpad **Doctoral Study Program in Nutritional Sciences IPB** University Tel.: (0251) 8622642 Fax:e-mail: pascasarjanagizi@apps.ipb.ac.id **Sponsors** Individual (Individual/Private/National grant/International grant) Clinical Monitor Dr. Lucky Angkawijaya Roring, M.Pd., AIFO Other Supervisors/Researchers: 1. Prof. Dr. Rimbawan 2. Prof. Dr. Ir. Hardinsyah, MS 3. Prof. Dr. Ir. Hadi Riyadi, MS Research Title: The Effect of a Balanced Nutritional Diet on Cardiovascular Risk Factors Among Two 3. Types of FTO Gene rs9939609 Obese Young Adult Women 4. Multicenter □Yes **Primary Research Center:** Satellite Research Flashlight: √ No 5. Study √ Not cooperation □National cooperation □International, number of countries please specify: □Involving a foreign Chief Researcher (attach permission, Institutional MoU, Researcher visa) 6. Filled in if a foreign research leader is involved No. Name, title, institution **Duties & Functions** Tel., Fax, HP, e-mail: of the foreign Research Chair 1. 2. 3. Research Place (Mention the name of the hospital, treatment room, polyclinic, or other health 7. service location): Screening of potential subjects, signing of the INFORMED CONSENT, collection of subject blood specimens, and data collection were carried out at the Health Services (Polyclinic), Universitas Pendidikan Indonesia Address: Jl. Dr. Setiabudhi No. 229, Isola, Sukasari, Bandung City The doctor responsible for examining the subject, taking samples and managing if any side effects occur: Dr Lucky Angkawijaya Roring, M.Pd., AIFO

| | | essary, collection of addi<br>ct's place if the subject p | | lete data | is carried out o | nline/by telephone or at th | e |
|---|---|---|---|---|---|---|---|
| | | specimen testing was ca<br>jaran University. | arried out at the | Molecula | r Genetics Labo | oratory, Faculty of Medicin | Э, |
| 8. | Resea | rch Time Plan: | | Starting: | November | Completed: February 202 | 4 |
| | ± 4 m | onths | | 2023 | | | |
| 9. | Data | Collection Time Starting: | November 2023 | to Februa | ary 2024 | | |
| 10. | Has T | his Protocol Been Submit | ted to Another I | Ethics Com | nmission? | | |
| | □Yes | | | | □Accepted | | |
| | | , attach a photocopy of t | he document! | - | □Rejected | | |
| | √ No | , | | | | | |
| 11. | | ation and Details of Resea | arch Funds (Hum | ıan Resoui | rces, Consumab | les, etc.): | |
| | No. | Type of Spending | | Compone | ent | Fee Required | |
| | 1 | Material | ATK | | | IDR 500,0 | 00 |
| | 2 | Material | Diet Procurem | ent (20x3x | (30x45,000) | IDR 81,000,0 | 00 |
| | 3 | Material | Elisa Kit (IL-6; | hs-CRP; a | adiponectin) | IDR 23,532,0 | 00 |
| | 4 | Material | DNA isolation | kit (40x200 | 0,000) | IDR 8,000,0 | 00 |
| | 5 | Material | Primary (1x400 | 0,000) | | IDR 400,0 | 00 |
| | 6 | Material | Primary Design | n Services | (1x150,000) | IDR 150,0 | 00 |
| | 7 | Material | Subject Rewar | d (40x35,0 | 000) | IDR 1,400,0 | 00 |
| | 8 | Data collection | FGD research | preparatio | on (5x105,000) | IDR 525,0 | 00 |
| | 9 | Data collection | Survey Office 40x8,000) | r's Honora | arium (Screeni | ng: IDR 320,0 | 00 |
| | 10 | Data collection | Temporary (40x18,000) | Blood | Glucose T | est IDR 720,0 | 00 |
| | 11 | Data collection | Researcher Ac | lministratio | on Honoraria | IDR 300,0 | 00 |
| | 12 | Data collection | Transport subj | ect + office | ers (43x25,000x | (2) IDR 2,150,0 | 00 |
| | 13 | Data collection | Data collection | meetings | (5x105,000) | IDR 525,0 | 00 |
| | 14 | Equipment Rental | Research Equi | ipment (2x | (350,000) | IDR 700,0 | 00 |
| | 15 | Specimen Analysis | PCR Gene Am | plification | (42x100,000) | IDR 4,200,0 | 00 |
| | 16 | Specimen Analysis | Sequencing (4 | 2x350,000 | )) + (42x10,000) | ) IDR 15,120,0 | 00 |
| | 17 | Specimen Analysis | Electrophoresi | s (42x50,0 | 000) | IDR 2,100,0 | 00 |
| | 18 | Specimen Analysis | Elisa Analysis | (3x1,800,0 | 000) | IDR 5,400,0 | 00 |
| | 19 | Data analysis | Honor Data Pr | | | IDR 1,540,0 | 00 |
| | 20 | Data analysis | Meeting Consu | umption Co | osts (5x105,000 | )) IDR 525,0 | 00 |
| | 21 | Reporting and Output | International S | eminar Fe | es | IDR 3,000,0 | 00 |
| | 22 | Reporting and Output | International S | cientific Pu | ublication Fees | IDR 3,500,0 | 00 |
| | | | Total | | | IDR 155 607 0 | nΩ |

### B. Clinical Trials

### Research methods

1. A summary of the research proposal includes the reason/motivation for conducting the research, the aims/objectives and benefits of the research, as well as the risks that may arise along with how to overcome them (written in language that is easy for non-doctors to understand):

Reason/Motivation for Conducting Research:

One nutritional strategy for obese individuals to lose weight is diet modification. Previous studies have shown that moderate weight loss (5–10% of initial body weight) achieved through lifestyle changes is associated with improvements in the cardiometabolic abnormalities characteristic of obesity (Espeland et al. 2007; Zomer et al. 2016). There have been studies and meta-

analyses that examine FTO gene polymorphisms coupled with certain types of dietary intervention which are then associated with changes in nutritional status, body composition, and various inflammatory and hormonal biomarkers in obese subjects (Razquin et al. 2010; De Luis et al. 2012b; De Luis et al. 2015a; De Luis et al. 2015b; Luglio et al. 2017; Di Renzo et al. 2018; De Luis et al. 2020; Parastouei et al. al. 2020), however, some things are still unclear and limited. Apart from that, no one has ever linked the FTO gene polymorphism to the Balanced Nutrition Diet intervention which is the reference in Indonesia, as well as its effect on cardiovascular risk.

### Research purposes:

### General purpose:

Examining the Effect of a Balanced Nutritional Diet on Cardiovascular Risk Factors Among Two Types of FTO rs9939609 Gene in Obese Young Women.

### Special purpose:

- 1. Analyze differences in the body composition of obese young women between A allele carriers (AC) and TT allele homozygous (TH) groups after Balanced Nutrition Diet intervention
- 2. Analyze differences in biomarkers of inflammation related to cardiovascular risk (interleukin (IL-6), high-sensitivity CRP (hs-CRP), and adiponectin (ADP)) of obese young women between A allele carriers (AC) and TT allele homozygous (TH) groups after Balanced Nutrition Diet intervention

### Benefits of research:

For research subjects, subjects can find out the allele type of the FTO rs9939609 gene themselves as an illustration of genes related to obesity and that can be used as a basis for precision nutrition interventions and will receive nutritional education about balanced nutrition. For the public, it is hoped that this research can increase knowledge about consumption recommendations, especially to normalize nutritional status and reduce the risk of cardiovascular disease by improving health status, especially for young adult women. For educational institutions, it is hoped that this research will provide new scientific evidence in the field of nutrigenomics regarding the interaction of genes and diet influencing the risk of obesity and cardiovascular disease. For the government, it is hoped that it can become a reference for making a policy to reduce obesity cases in Indonesia.

### Number of Research Subjects:

This research uses a hypothesis testing formula for 2 independent samples based on Sastroasmoro & Ismael (2014):

$$n_{=}n_{2}=2\left[\frac{(Z_{a}+Z_{b})S}{X_{1}-X_{2}}\right]^{2}$$

The results of calculations using data from previous research (De Luis et al. 2015b) resulted in 7 people. This study used 4 groups, namely 2 control groups and 2 intervention groups, adding an anticipated dropout of 50%, the total number of subjects was at least 44 people or 11 people per group.

### Information:

n = minimum number of subjects

 $Z\alpha$  = type I error (1.96)

Zb = type II error (1.28; power 90)

S = standard deviation of the two groups

X1 – X2 = desired clinical difference (difference in weight between Allele T and Allele A)

Research by De Luis et al. (2015b) is a consideration for the expected weight loss of subjects in this study, namely assuming a weight loss of  $\pm 1$  kg in A allele carriers and  $\pm 0.35$  kg in homozygous T subjects after 1 month of intervention with the balanced nutritional diet provided.

How to Choose Research Subjects

Inclusion Criteria: 1) Obese women (body fat percentage >35%) who have light physical activity based on PAL (can select prospective subjects who have participated in preliminary research to completion); 2) Sundanese ethnicity (father, mother, grandfather, grandmother originally from West Java); 3) normal fasting blood pressure and blood sugar; 4) aged 18-25 years (based on Loos and Yeo (2014) that the relationship between the FTO gene and obesity is greatest in young adulthood); 5) not currently pregnant or breastfeeding; 6) willing to participate and sign informed consent. Exclusion Criteria: 1) currently pregnant and breastfeeding; 2) have a history of chronic disease; 3) regularly consume antioxidant supplements and/or phytopharmaceuticals; 4) currently participating in other research. Risks that may arise and how to overcome them: Potential harm to the procedure being performed is very rare. The potential that may be encountered is limited to conditions of infection and the formation of hematomas (blood clots due to needle sticks). This risk can be reduced by treatment by experienced professionals and the use of disposable equipment and aseptic procedures, as well as appropriately sized needles to minimize the occurrence of hematomas. Apart from that, there may be a danger of bacterial contamination from intervention foods made by researchers. This can be prevented by maintaining hygiene and sanitation during preparation, processing, packaging, and when providing intervention food. In addition, the possibility of side effects or dangers from consuming the dietary intervention provided is prevented by collecting data on dietary restrictions/allergies for each subject before the intervention is carried out. Research Methods (There may be more than one) √ Randomization 2. √ Open labelled □Placebo □Cross-over √ Treatment controlled √ Parallel ☐Single Blind □Double Blinds □Others mentioned, 3. New Drug Research (Investigational New Group=IND)/New Equipment (Investigational New Equipment =INE)/New methods or techniques: □Ther DINE √ There Health isn't any e are: Reg No. POM: Reg No. POM: Department Name: Name: Permit: ☐There is Sponsor: Company name: Sponsor: Company name: □No If there is, attach it Information About Try Ingredients: a. Efficacy: b. Security: -4. For Genetic Research, Indicate Whether Genetic Engineering Techniques Are Used: √ No: ☐Yes, it has been reviewed ☐Recombinant DNA Advisory Committee ☐Biosafety Committee 5. This data is filled in if it concerns clinical drug Companion Medicine Drugs Tested trials Generic name: a. b. Trade name: c. Chemical name:

| | d. | Pharmacol | ogy class: | | |
|---|---|---|---|---|---|
| | e. | Dosage for | m and drug strength: | | |
| | f. | Packaging: | | | |
| | g. | Way of giv | ing: | | |
| | h. | Expired da | te: | | |
| | i. | Batch Num | nber: | | |
| | j. | Analysis ce | ertificate: | | |
| | k. | CPOB Cert | ificate: | | |
| | I. | Type and o imported: | quantity of medicines to be | | |
| | m. | Manufactu | irer's name and address: | | |
| | n. | - | name and address: | | |
| | 0. | | n status of the test drug in<br>htries (if any, please attach | | |
| | | it) | | | |
| | p. | | al phase: Phase I Phase II | | |
| 6. | How to Go | et Research | ☐Individual contacts V Ba☐Reference☐Advertisem | | |
| 7. | Subject Co | riteria: | | <u> </u> | |
| | □Prone | to | □Child's age < 12 years □Prisoner □People with impaired cogs □Pregnant mother □TNI and Police □Others, please specify: | | usness<br> |
| | √ Not Vu | ılnerable | | | |
| 8. | carried ou<br>Reference | ıt, data on s | inical trial using human subje<br>afety and efficacy from previo<br>tle, Journal): –<br>Results: – | | |
| | been carr<br>Reference<br>Salimei P<br>compositi<br>12. doi:10<br>Resume o<br>the Medit<br>Mediterra<br>of FTO are | ied out, safe<br>es (Name, Ti<br>, De Lorenz<br>ion and weig<br>0.1186/s129<br>of Research l<br>terranean di<br>anean Diet is<br>e still uncert | own or others) of the action ety and efficacy data from presitle, Journal): Di Renzo L, Cioco A. 2018. Influence of FTG et al. 2018. Influence of FTG et al. 2018. Influence of FTG et al. 2018-1680-7. Results: Randomized clinical et al. 2018-1680 et al. 2018-168 | vious studies/in other couccoloni G, Falco S, Abenav<br>O rs9939609 and Medite<br>al trial NCT01890070 NCT.<br>trial examining the effects<br>weight loss. The results of | untries): V No□Yes voli L, Moia A, Sinibaldi erranean diet on body I J Transl Med. 16(1):1– s of FTO rs9939609 and obtained show that the |
| 9. | | ial Process | nistration (dosa ragiman in | vacive and non investive a | rocoduros comparisos |
| | drugs, | placebo):<br>Following ir | nistration (dose regimen, inv<br>nformed consent and initial so<br>nts to establish baseline data. | creening, blood samples w | vill be collected from all |

be conducted using the block randomization method, based on the FTO gene allele. This process will involve two sample randomization blocks: one for A carriers allele and another for T homozygous individuals. Each block will then be randomized and divided into two groups, maintaining a 1:1 ratio between control and dietary intervention. Following randomization, four groups will be formed: two groups receiving the Balanced Nutrition Diet intervention (DAC: A allele carriers + Diet; and DTH: homozygous T allele + Diet), and two control groups (CAC: A allele carriers; and CTH: homozygous T allele). Nutrition education will be provided to all groups. The intervention period will span 4 weeks (28 days), after which a second blood draw will be conducted to gather endline data.

The Balanced Nutrition Diet is meticulously designed to supply the body with nutrients in suitable types and quantities, adhering to the principles of food diversity which include variety, balanced proportions, correct amounts, and consistency. Additionally, it emphasizes the "Fill My Plate" guideline, advocating for the consumption of all five food groups daily or at each meal. Portion sizes of the Balanced Nutrition Diet are structured according to the "Balanced Nutrition Tumpeng" model, encompassing 3-4 portions/day of carbohydrates, 2-3 servings/day of fruit, 3-4 servings/day of vegetables, and 2-4 servings/day of side dishes, with restrictions set at 4 tablespoons of sugar, 1 teaspoon of salt, and 5 tablespoons of oil per day, alongside a recommendation of drinking 8 glasses of water daily.

During the intervention period, food is provided three times a day - breakfast, lunch, and dinner - following a 28-day menu cycle. The researcher bears the sole responsibility for covering the cost of all food provided to the intervention group during this 28-day period. The Balanced Nutrition Diet offered adheres to specific macronutrient distribution ratios of 45-55% carbohydrates, 15-20% protein, and 20-25% fat, as outlined by Almatsier (2010). Complex carbohydrates, such as whole grains, are prioritized, while protein sources lean towards low-fat options, with half derived from plant-based sources. Monounsaturated and polyunsaturated fats are favored, and organic ingredients are preferred whenever possible.

Each meal's composition adheres to the "Fill My Plate" principle, and daily portions follow the "Balanced Nutrition Tumpeng" concept. Specifically, the diet provided by Eat & Fit Catering adheres to certain guidelines, including cooking methods that eschew fire and oil frying in favor of boiling, sautéing, or roasting techniques. Canola oil is the preferred oil, sodium-reduced salt is utilized, and mushroom stock serves as the primary flavouring agent, ensuring both healthfulness and taste. For each subject, energy requirements were calculated according to resting energy expenditure (REE) estimates using Mifflin-St. Jeor Equation (Mifflin et al. 1990). REE is then multiplied by the physical activity level (PAL) according to WHO-FAO that has been obtained.

### REE (women)= $(9.99 \times Body Weight) + (6.25 \times Height) + (5 \times Age) - 161$

The dietary distribution to subjects occurs three times, facilitated by couriers from the catering party. Should the delivery fall beyond the catering courier's radius, online delivery services will be utilized, with costs borne by the researcher.

In contrast, the control group subjects do not adhere to a specific diet regimen. However, they will receive general guidance on healthy eating habits and will be monitored closely. Nonetheless, their energy requirements will still be assessed based on REE and physical activity levels, as previously mentioned.

### b) Determination of outcome indicators:

Evidence shows that compared with TT wild type, the risk allele A FTO rs9939609 showed significantly higher body weight, body mass index, waist circumference, hip circumference, and waist-to-hip ratio (Mangge et al. 2011; Tupikowska-Marzec et al. al. 2019; Mehrdad et al. According to Chrostowska et al. (2013), evidence is growing that the waist-hip circumference ratio is a stronger indicator of cardiovascular disease than body mass index. The meta-analysis of Gholamalizadeh et al. (2020), showed that carriers of the A allele of the FTO rs9939609 polymorphism had a higher fat percentage. The research results of Dorling et al. (2021) showed

the FTO SNP rs9939609 was associated with changes in REE adjusted for fat mass and lean mass, with the AA allele showing a decrease compared to TT.

Several studies have been conducted looking at the relationship between the FTO rs9939609 genotype and interleukin-6 (IL-6) levels, but only a few have shown real differences (de Luis et al. 2012b; Zimmermann et al. 2011; de Luis et al. 2016; Magno et al. al. 2018; Hosseini et al. Studies have also been conducted that there is an association of FTO rs9939609 with higher levels of C reactive protein (CRP) (Fisher et al. 2009; Sun et al. 2010; Lappalainen et al. 2011; Tupikowska-Marzec et al. 2019). However, other studies show contradictions (Zimmermann et al. 2011).

Research by Mehrdad et al. (2020a) showed that subjects with A allele carriers (AA and AT) had lower adiponectin levels than wild-type subjects (homozygous TT) with homozygous AA allele types having the lowest values although not significantly different. Several other studies also show the same thing in both obese and other types of adult subjects (Saucedo et al. 2017; Isgin-Atici et al. 2021). However, research by de Luis et al. (2016) and Duicu et al. (2016) showed a contrast, namely that adiponectin levels were lower in the TT genotype group compared to the AA genotype group. Based on what has been explained above, several outcome indicators that will be analyzed are waist-hip circumference, mass and total fat percentage &visceral, interleukin-6 levels, hs-CRP levels, and adiponectin levels.

### Statistical analysis

The data obtained were tested statistically using SPSS statistical software for Windows (IBM version 26.0, SPSS Inc., Chicago, III., USA). The normality of variable distribution was verified with the Shapiro-Wilk test. Analysis of Variance (ANOVA) was used for all baseline data. Paired samples t-test was used to see changes in calorie intake, macronutrients, BW, BMI, waist circumference, hip circumference, waist-hip ratio, RM, percent total fat, visceral fat, subcutaneous fat, skeletal muscle, IL-6, hs-CRP, and adiponectin between before and after intervention. Data are presented as mean  $\pm$  SD and P < 0.05 was considered statistically significant.

- c) Planned interim analysis: There is no interim analysis in this study.
- d) Clinical trial termination procedures: Referring to the guidelines for good clinical trials in Indonesia (POM RI 2016), clinical trials are terminated if clinical trial safety problems occur, such as serious undesirable events and serious side effects of the test product. The principal investigator will report the KTDS to the ethics committee no later than 3 days after the incident is discovered. The possibility of KTDS that could occur in this study is that the patient requires hospital treatment as a result of the intervention process.
- e) Estimated research time required for one subject per procedure: ±4 weeks
- f) Ethical issues (state your opinion about the ethical issues this research may encounter):
  - Respect for person (respect for human dignity):
     Subjects in this study took part based on their own conscious choice, there was no element of coercion.
    - Subjects have the right to be protected, including that all Subject data will be kept confidential.
  - Beneficence(beneficial) Non-maleficence (not harmful):
    - This research optimizes benefits and minimizes harm to subjects.
    - The results of the research will be useful for society.
    - The research design has been made as clear as possible.
    - Researchers have competencies that are appropriate to the research topic to be conducted.
  - Justice(justice):
    - Subjects are treated the same/or there is no differentiation between subjects.

### There is no conflict of interest

- 10. Adverse Event reporting plan(AE)
  - Recording (What will be reported): Each incident must be recorded in detail regarding the time it occurred and the causes to avoid similar incidents and as additional data for research progress reports.
  - b. Analysis and action procedure:
    - 1. Anthropometric Measurements

After an overnight fast for 12 hours, all subjects underwent anthropometric evaluation. All individuals were instructed to remove their shoes and wear as light clothing as possible before undergoing measurements. Body weight, mass & percent body fat were measured with a Bioelectrical Impedance Analyzer (BIA). Body height was evaluated using a stadiometer to the nearest 0.1 cm. BMI is calculated using the formula = body weight/height2 (kg/m2). Waist circumference and hip circumference were assessed using a flexible steel metric tape to the nearest 0.5 cm. The waist-to-hip ratio (WHR) was analyzed and evaluated according to clinical risk thresholds, equivalent to WHR > 0.9 for men and WHR > 0.85 for women.

### 2. Blood Sample Analysis

A venous blood sample of around 6-10 cc is taken using a sterile syringe by competent licensed medical personnel. The blood is then divided into two different sterile tubes (Vacutainer®). The first tube is a purple cap tube containing EDTA, while the second tube is a yellow cap tube containing separator gel. After that, the sample is put on ice to be immediately taken to the testing site. The samples in the purple tube will then be processed for DNA and RNA isolation. DNA isolates were used for analysis of FTO gene variants using PCR and sequencing. Blood samples in yellow tubes were used for analysis of serum levels of interleukin-6, hs-CRP, and adiponectin using the ELISA method. All blood analyzes will be carried out at the Molecular Genetics Laboratory, FK UNPAD. The remaining samples were stored at -80 °C to be retested if necessary.

- c. Emergency request system: Each subject will be given a contact for researchers and doctors who can be contacted if there are complaints of illness related to the intervention. Researchers and doctors can be contacted 24 hours during the research period regarding interventions for emergency response preparedness. If there is an emergency, the subject will be taken to the emergency room at Hasan Sadikin Hospital.
- d. Termination of subjects in research due to adverse events: If an undesirable event occurs, it must be immediately reported to the researcher. Researchers will then coordinate with parties who feel it is necessary to carry out follow-up as soon as possible. Then the researcher will assess whether the subject needs to be discontinued in the study after consulting with a clinical trial expert.
- 11. If this research uses human subjects, are the costs of dealing with side effects the responsibility of this research? ☐No ∨ Yes
  - If yes, post-research responsibilities (capacity building, benefits to local community, continuation of therapy on the subject, etc.)
  - Is the subject insured? √ No□Yes

If "yes" please state the insurance institution: —
Duration of Insurance and/or responsibility of the researcher towards the subject? —

12. If we use biological samples, will they be sent overseas? √ No ☐Yes, please state the destination country and attach itdrafts *Material Transfer Agreement* (MTA)!

| <u> </u> | PIU | cess of Obtain | ilig Approval Arter Exp | nanation ( | INFORIVIED | COI | N3EN 1 | ieu Conse | ent (ic) |
|---|---|---|---|---|---|---|---|---|---|
| 1. | Ехр | lained(There m | MED CONSENT IS nay be more than | lIndividua | ٧ | Grou | ıp | □Guar | dian |
| | one | answer): | | | | | | | |
| 2. | a. | Who explain | ıs? | ı | Principal Researcher | | | | |
| | b. | When will it | be explained? | | Before INFORMED CONSENT | | | | |
| | | | | 9 | screening and signing is carried out | | | | |
| | c. | Are subjects | given enough time to | make a d | ecision? | ١ | ⁄es | | |
| | d. | Who signed | the INFORMED CONSI | ENT? | | | The prospectiv | e subject | itself |
| | e. | Who witness | sed the INFORMED CC | ONSENT sig | ning? | tant | | | |
| | | | | | | ( | doctor/nurse/ | /midwife <sub>/</sub> | /nutritionist |
| | | | | | | ) | | | |
| 3. | Eth | | hat the subject may fa | ace | | | | | |
| | a. | Research risl | | | | | | ı | |
| | | | outine health service | | | | lYes | | No |
| | | + | de effects on the subje | | | lYes | | No | |
| | | 3. Contrary t | to norms and customs | | | | lYes | ٧ | No |
| | | | losses and stigmatizat | | | lYes | ٧ | No | |
| | | subject | | | | | | | |
| | b. | Benefits of t | aking part | | | | | | |
| | | | vledge increases | | | ٧ | Yes | | □No |
| | | 2. Get health | n services | | | √ Yes | | | □No |
| | | 3. Incentives | 5 | | | | lCash□No | | |
| | | | | | | ٧ | Goods/Souve | nirs | |
| | | 4. Compensa | ation | | | | lInsurance √ C | ash | |
| | | | | | | | lNo□Etc | | |
| | c. | | fluence (coercion) | | | | | | |
| | | | nip between Chief Res | 1 | | | No | □The | |
| | | 2. If there | □Doctor-patient | | er/lecturer | - | □Superiors | | □Etc |
| | | is: | | pupils/st | | | subordinate | | |
| | d. | If the study uses healthy people, explain how the health checks will be carried out: | | | | | | | |
| | | • If the stud | dv uses sick people. ex | to diagnos | se and name the doctor responsible! | | | | |
| | | | s study used young ad | • | - | | | • | |
| | | | d by a nutritionist bas | | • | | | _ | , |
| | | | ole doctor: dr. Lucky A | | | | • | | |
| | | Кезропзік | The doctor. ar. Lucky A | iigkawijay | a Norma, N | vi.r u. | , All O. (00112 | 220137). | • |
| D. | E:11 | in the Consent | t Information After Ex | nlanation | /INIEODNIE | ED C | DNISENIT\/Info | rmad Car | acont (IC) |
| 1. | | | Agreement After the | • | • | | | illeu Coi | isent (ic) |
| 1. | | | nary information | Jubject Lx | V Yes | LXPIC | | | |
| | | | applied to the subject | , | v res<br>√ Yes | | □No | □Not Av | zailahla |
| | | Benefits for the | | , | √ Yes | | □No | □Not A | |
| | | | • | | √ Yes | | □No | □Not A | |
| | | Potential dange | <u>= </u> | | | | □No | | |
| | | Right to resign | | | √ Yes | | □No | □Not A | |
| | | ncentives for s | • | | √ Yes | | | | |
| | | Type of incention | • | | √ Yes | | □No | □Not A | |
| | n. ( | Compensation ' | tor subjects | √ Yes | | □No | □Not A | valiable | |

| 2. | Specimen Collection (Statements 2b-2d are filled in if the a answer to 2e is "yes") | answ | er to 2a is "yes" an | nd 2f-2g if the |
|---|---|---|---|---|
| | a. Was a specimen taken from the subject? | | □No | √ Yes, Blood |
| | b. Is there information on the number of specimens taken | 1? | √ Yes | □No |
| | $c. \ \ $ Is there any information about the frequency of collection | on? | √ Yes | □No |
| | d. Is there any information about how to collect it? | | √ Yes | □No |
| | e. Was there any invasive procedure on the subject? | | √ No | ☐Yes, Name it |
| | f. Is there any information about the potential risks of taking? | | √ Yes | □No |
| | g. Is there information about how to handle risk-taking? | | √ Yes | □No |
| 3. | Subject Confidentiality | | | |
| | a. Is there any information about subject | ۷ Ye | S | □No |
| | confidentiality? | | | |
| | b. Is there any information about specimen | √ Ye | S | □No |
| | confidentiality? | | | |
| | c. Is there any information about data confidentiality? | √ Ye | S | □No |
| 4. | Contact person local for respondents, please specify: Putri | Novi | tasari (081122272 | .91) |
| | Contact person centre for respondents, please specify: Put | tri No | vitasari (0811 <mark>2227</mark> | 7291) |

### E. Statement

| 1. | priva | he head of research been involved/punished for criminal/disciplinary action by the public or a te medical organization/an authorized body? ☐Yes, explain |
|---|---|---|
| 2. | | long will research data be kept by the Principal Researcher? 1 to 2 years after the research is pleted |
| 3. | What | precautions are taken to maintain the confidentiality of health data? |
| | ٧ | Research documents/files will be stored in a secure location and can only be accessed by officers involved in the research |
| | ٧ | Computer data is only intended for officers involved in research and can be accessed using passwords and personal access |
| | ٧ | Before accessing any research-related information, personnel must sign a consent form to protect the security and confidentiality of the subject's health information |
| | <b>\</b> | Before opening research files, officers must sign an agreement to maintain the confidentiality of the documents |
| | ٧ | Where possible, identification of research subjects is removed (anonymous) from information related to research |
| | | Others, explain |
| 4. | | be responsible for filling out this form and will carry it out in accordance with the proposed arch proposal and in accordance with the principles of research ethics. |



### RESEARCH ETHICS COMMITTEE JI. Prof. Eijkman No. 38 Bandung 40161 Telp. & Fax. 022-2038697, website: kep.unpad.ac.id, email-sekretariat: kep@unpad.ac.id

Bogor, 05 Juni 2023

Penelit Utama,

Mengetahui,

Ka. Departemen/Prodi

Dr. Drs. Rimbawan

Putri Novitasari, S.Gz., M.Si

Pembimbing I,

Dr. Drs. Rimbawan

Pembimbing II,

Prof. Dr. Ir. Hardinsyah, M.S.

Pembimbing III

Prof. Dr. Ir. Hadi Riyadi, M.S.

### **INFORMATION SHEET**

### The Effect of a Balanced Nutritional Diet on Cardiovascular Risk Factors Among Two Types of FTO Gene rs9939609 ini Obese Young Women

I am Putri Novitasari, a Doctoral (S3) student in Nutrition Science from the IPB University who is conducting research for her dissertation. I invite you to participate in this research, your participation in this research is voluntary, so you can decide whether to participate or not.

### **Research purposes:**

The general aim of this research is to

Examining the Effect of a Balanced Nutritional Diet on Cardiovascular Risk Factors Among Two Types of FTO Gene rs9939609 in Obese Young Women.

Meanwhile, the specific aim of this research is to

- 1. Analyze differences in the body composition of obese young women between A allele carriers (AC) and TT allele homozygous (TH) groups after Balanced Nutrition Diet intervention
- 2. Analyze differences in biomarkers of inflammation related to cardiovascular risk (interleukin (IL-6), high-sensitivity CRP (hs-CRP), and adiponectin (ADP)) of obese young women between A allele carriers (AC) and TT allele homozygous (TH) groups after Balanced Nutrition Diet intervention

### Why Subject was chosen:

You were selected for this study because you meet all the inclusion criteria, namely: 1) Have a fat percentage of >35% and have light physical activity based on PAL (and have participated in preliminary research to completion); 2) Sundanese ethnicity; 3) normal fasting blood pressure and blood sugar; 4) aged 18-25 years (based on Loos and Yeo (2014) that the relationship between the FTO gene and obesity is greatest in young adulthood); 5) not currently pregnant or breastfeeding; 6) willing to participate and sign informed consent.

### **Procedures/Procedures:**

You will be invited to the UPT Health Services, Indonesian Education University gathered with other respondents at one time. First of all, an explanation of the aims and objectives of the research is provided, followed by an explanation of the actions/treatment that will be carried out in this research including the benefits and disadvantages of being a research subject including the compensation you will receive and the right to withdraw from the research. Then there will be a distribution of informed consent and if the prospective subject is willing and signs the informed consent and passes the screening, they will officially become research subjects.

The first stage of screening is assessment, physical examination (blood pressure, pulse and fasting blood sugar), and anthropometry (body weight, height, waist circumference and hip circumference, total & abdominal fat mass and percentage) as basic measurements for internal screening All prospective subjects had fasted overnight. If you do not pass the screening, then you will be declared disqualified. On the other hand, if you pass the screening then you are declared a research subject. Medical assessments including blood pressure and blood sugar checks by nurses/midwives and health checks by doctors are evaluated before and after the intervention.

Screening of potential subjects, signing of the INFORMED CONSENT, collection of subject blood specimens, and data collection were carried out at the UPT Health Services (Poliklinik), Indonesian Education University. Address: Jl. Dr. Setiabudhi No. 229, Isola, Sukasari, Bandung City

After that, on the same day, you will have a blood sample taken as initial biochemical data. After the initial biochemical data was obtained, samples were randomized using the block randomization method based on the FTO gene allele. There will be 2 sample randomization blocks, namely the A carriers allele block, and the T homozygous block. Each block was randomized and divided into 2 groups with a ratio of control to dietary intervention (1:1). Because this research uses a parallel design, you only experience one type of intervention. Randomization was carried out using a roll of paper containing subject codes without replacement. Randomization was carried out by personnel who did not participate in research activities. After that, they enter the intervention stage for 4 weeks (28 days) according to the group. After 4 weeks (28 days), a second blood draw will be taken as final biochemical data. Analysis of the FTO gene and other blood biochemistry will be carried out at the Molecular Genetics Laboratory, Faculty of Medicine, Padjadjaran University.

Height measurement uses a microtome with an accuracy of 0.1 cm, BB measurement uses a step scale with an accuracy of 0.1 kg. Waist circumference and hip circumference were measured using a body circumference meter with an accuracy of 0.1 cm. Mass and percentage of total & visceral fat using the Bioelectrical Impedance Analyzer (BIA) with an accuracy of ± 400 grams for a body weight of 0.0–40.0 kg, while for a body weight of 40.0–135.0 kg, the accuracy is ± 1%. Blood biochemical data include high sensitivity-C-reactive protein (hs-CRP); interleukin-6 (IL-6), and plasma adiponectin. Gene data examined includes FTO gene variations. Consumption data includes: recording food consumption (self-administered food record). Food records 2x24 hours were carried out before the intervention started and during the intervention. Subjects will be instructed to record or record the type and weight of food and drinks consumed and then the nutrients will be reviewed and calculated. Compliance with the consumption of a Balanced Nutrition Diet using Googleform which must be filled in by the intervention group every day. The minimum limit for subject compliance is 80% of the entire diet provided. Physical activity data includes the length of time doing various types of physical activity within 24 hours, used to estimate the subject's energy expenditure.

Food was provided during the intervention period 3 (three) times each day, namely breakfast, lunch and dinner. The food menu uses a 28-day menu cycle. The cost of all food provided to the intervention group during the 28 days was the sole responsibility of the researcher.

The characteristics of the Balanced Nutrition Diet that will be provided have a distribution of the composition of the macronutrients that will be intervened in are as follows: 45-55% carbohydrates, 15-20% protein, and 20-25% fat (Ministry of Health 2014). The type of diet and portions that will be given are the same for each feeding unless there are certain food restrictions or allergies, the type of food will be adjusted specifically to that individual. The calories that will be given range from 300-400 Cal for breakfast, 400-500 Cal for lunch, and 300-500 Cal for dinner.

The choice of carbohydrates should be varied and should be complex carbohydrates such as whole grains. The choice of protein type is prioritized from low-fat protein sources and half of it is vegetable protein. The choice of type of fat is prioritized in the form of monounsaturated and polyunsaturated fats. If possible, food ingredients should be prioritized in the form of organic food. The composition of each meal refers to the principle of "Fill My Plate" and the daily portion refers to the principle of "Balanced Nutrition Tumpeng". The characteristics of the diet that will be provided specifically from the Eat & Fit Catering diet consist of 1) Cooking methods that use boiling/sautéing/roasting techniques without fire and avoiding frying techniques

with oil; 2) The oil used is canola oil; 3) The salt used is a special type of salt which has less sodium content; 4) The flavouring used is mushroom stock.

For each subject, energy requirements were calculated according to resting energy expenditure (REE) estimates using Mifflin-St. Jeor Equation (Mifflin et al. 1990). REE is then multiplied by the physical activity level (PAL) according to WHO-FAO that has been obtained.

### REE (women)= (9.99 x Body Weight) + (6.25 x Height) + (5 x Age) - 161

The technical distribution of diets to subjects is delivered 3 times by couriers from the catering party. If the delivery is outside the delivery radius of the catering courier, the food will be delivered by online delivery services and costs will be charged to the researcher.

In contrast, in the control group, subjects do not follow a specific diet, but they will also receive general recommendations about healthy eating habits and will only be monitored, however, their energy needs will still be evaluated based on REE and physical activity as mentioned above.

### **Risks and inconveniences:**

The risks in this study are very small/minimal, but there is inconvenience because your time will be taken up for collecting data and recording dietary compliance (for those in the intervention group). Apart from that, the potential that may be encountered is limited to conditions of infection and the formation of hematomas (blood clots due to needle sticks). This risk can be reduced by treatment by experienced professionals and the use of disposable equipment and aseptic procedures, as well as appropriately sized needles to minimize the occurrence of hematomas. Apart from that, there may be a danger of bacterial contamination from intervention foods made by researchers. This can be prevented by maintaining hygiene and sanitation during preparation, processing, packaging, and when providing intervention food. In addition, the possibility of side effects or dangers from consuming the dietary intervention provided is prevented by collecting data on dietary restrictions/allergies for each subject before the intervention is carried out.

### Benefits (direct to the subject and general):

For you, you can find out the allele type of the FTO rs9939609 gene as an illustration of genes related to obesity and which can be used as a basis for precision nutritional interventions and will receive nutritional education about balanced nutrition. For the public, it is hoped that this research can increase knowledge about consumption recommendations, especially to normalize nutritional status and reduce the risk of cardiovascular disease by improving health status, especially for young adult women.

### Alternative procedure:

"There isn't any"

### Data confidentiality:

Researchers will guarantee the confidentiality of research data.

### Estimated number of subjects to be included:

The total number of research subjects who will take part in this research is around 44 people.

### Volunteerism:

Subject participation is voluntary without any coercion and is accompanied by responsibility until the completion of the research.

### **Subject Participation Period:**

You will be involved in the entire series of this research for approximately 2 months, consisting of 1 month intervention period and an additional 2 weeks each before and after the intervention period for preparation.

### Subjects can be excluded/withdrawn from research:

Drop-Out Criteria are 1) you state that you do not wish to continue; 2) indications of exclusion criteria were found in you during the research; 3) You did not undergo complete blood and/or other necessary tests.

### Possible funding from health insurance companies or researchers:

"no insurance was provided in this study"

### Incentives and compensation:

Transport costs when you go to the screening site and sign the INFORMED CONSENT will be reimbursed in cash amounting to IDR. 50,000,-. Those who have participated until the final data collection will be given incentives in the form of contact materials in the form of boxes and cutlery.

### Question:

If anything is unclear or you need to ask questions, please contact the principal investigator:

Putri Novitasari (08112227291): D Amerta Residence Jl. Pandanus III Block E1 No. 30 Bojongsoang District, Bandung Regency

Contact a doctor if any side effects occur: Dr. Lucky Angkawijaya Roring, M.Pd., AIFO

### APPROVAL AFTER EXPLANATION (INFORMED CONSENT) TO PARTICIPATE IN RESEARCH (INFORMED CONSENT)

I have read or received an explanation, am fully aware, understand and comprehend the objectives, benefits and risks that may arise in the research, and have been allowed to ask questions and have been answered satisfactorily, and can withdraw from participation at any time. then I agree/disagree\*) take part in this research, entitled:

### The Effect of a Balanced Nutritional Diet on Cardiovascular Risk Factors Among Two Types of FTO Gene rs9939609 in Obese Young Women

I voluntarily chose to take part in this research without pressure/coercion from anyone. I will be given a copy of the explanation sheet and the signed consent form for my records.

I agree: Yes No\*)

| | Date: | Signature (if not available, thumbprint can be used) |
|---|---|---|
| Participant Name: | | |
| Age: | | |
| Address: | | |
| Researcher Name: | | |
| Witness Name: | | |

<sup>\*)</sup> cross the unnecessary ones

### **CASE REPORT FORM**

### Case Report Form is available at: <a href="https://forms.gle/zscvmfcFvAzZJ6HcA">https://forms.gle/zscvmFcFvAzZJ6HcA</a>

| 7/20/23, 2:43 PM | | Case Report Form | 7/20/23, 2:43 PM | | | | Case Report Form | |
|---|---|---|---|---|---|---|---|---|
| | | | 5. | Pemeriksa | an Keseh | atan * | | |
| ( | Case Report Form | | | Mark only o | ne oval per | row. | | |
| P | Pengaruh Diet Gizi Seimbang terhadap Faktor | | | | Normal | Abnormal | | |
| | disiko Kardiovaskular pada Dua Tipe Gen FTO i | rs9939609 Wanita Dewasa Muda Obese | | Tekanan<br>Darah | 0 | 0 | | |
| 1. | Email * | | | Denyut<br>Nadi | 0 | 0 | | |
| | | | | Suhu | $\circ$ | | | |
| 2. | Nomor Subjek | | | Gula<br>Darah<br>Puasa | 0 | 0 | | |
| | Penapisan (Screening) | | | | | | | |
| 3. | Tanggal persetujuan informed consent * | | | | | | | |
| | Example: January 7, 2019 | - | | | | | | |
| 4. | Tanggal Penapisan | | | | | | | |
| | Example: January 7, 2019 | - | | | | | | |
| https://docs.googl | ie comformald/LJ2_leac1nKYFKPfb/seDO-jGeAE1a8cfeaE53c | cOWIZVOledtifresponses 1 | 1/5 https://docs.goog | le.com/forma/d/1. | J2_leac1nKYF | KP8zkeDO-jQeAE | alicheli 93cOWZ/GleditiFesponses | 2/5 |

| 7/20/23, 2:43 PM | | | | Case Report Form | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| 8. | Eksklusi * | | | | | | | | | |
| | Check all that ap | nlv | | | | | | | | |
| | Officer as that ap | | | | | | | | | |
| | | Ya | Tidak | | | | | | | |
| | Sedang hamil | | | | | | | | | |
| | dan<br>menyusui? | | | | | | | | | |
| | Memiliki | | | | | | | | | |
| | riwayat<br>penyakit | | | | | | | | | |
| | kronis? | | | | | | | | | |
| | Rutin | | | | | | | | | |
| | konsumsi<br>suplemen | | | | | | | | | |
| | atau obat- | | | | | | | | | |
| | obatan | | | | | | | | | |
| | fitofarmaka? | | | | | | | | | |
| | Sedang | | | | | | | | | |
| | berpartisipasi | | _ | | | | | | | |
| | pada | | | | | | | | | |
| | penelitian<br>lain? | | | | | | | | | |
| | | This conti | int is neither o | rested nor endorsed by Google. | | | | | | |
| | | | Goo | gle Forms | | | | | | |
| | | | | , | | | | | | |
| Https://docs.google | le com/formeld/1.12_leac | 1nKYFKPBelo | :00-j0sAE1s8 | des ESSONYES VIVES Bresponses | 55 | | | | | |
| | la comformald*1J2_leac | 1niCYFiCPBalu | sOO-jQeAE1s8s | | 55 | | | | | |
| Https://focs.google<br>750023, 2-43 PM | le constormald*132_leac | 1niCYFICPBcba | 00-j0+AE1+80 | бы:E33cOWZvOed8#нарогиня<br>Сана Парот Гот | 55 | 7/20/29, 2×3 PM | | | | Case Report Form |
| 7/20/23, 2:43 PM | a comformal/31,12_leac | 1:nKCYFIKPBeke | oDO-JORAE1888 | | 55 | | Inklusi * | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * | | oDO-jOeAE1e8e | | 55 | | Inklusi * | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow | al per row. | 000-j0#AE1#8 | | 55 | | | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow | | 000-j0eA81e8 | | 55 | | Inklusi * | Ya | Tidak | Ceas Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow | al per row. | 00-j0eAč1e6 | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 | Ya | Tidak | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow N BB aktual | al per row. | 000-j0eAE1e8 | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ov | al per row. | oDO-JORAE1s8 | | 55 | | Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak | Ya | Tidak | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow N BB aktual TB aktual | il per row. | oDO-jGeAE1e8 | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow N BB aktual TB aktual IMT | al per row. | oDO-jūeAE1e6e | | 55 | | Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow N BB aktual TB aktual IMT Total | il per row. | oo-joraliteb | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m² dan persen lemak >35%)? Etnis Sunda? | | | Class Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen | il per row. | oco-jos-Ačtso | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow N BB aktual TB aktual IMT Total | al per row. | OO-JORAETe6 | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m² dan persen lemak >35%)? Etnis Sunda? | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh | al per row. | oDO-jūrAĒ1ebe | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen | al per row. | oco-joražiteče | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah | | | Ceas Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow N BB aktual TB aktual IMT Total persen lemak tubuh Persen | al per row. | oco-joeAE1a6 | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen | al per row. | oco-josAžitso | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow N BB aktual TB aktual IMT Total persen lemak tubuh Persen lemak visoeral | al per row. | oco-joeAčtso | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark enly one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen lemak visceral Total massa | al per row. | oDO-jūeAE1ebe | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen lemak visceral Total Total persen | al per row. | oco-joeAE1a6e | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Cess Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark enly one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen lemak visceral Total massa | al per row. | oco-joealitelo | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen lemak visceral Total massa lemak tubuh Massa | al per row. | iOO-jOsAEtsio | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Class Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Total massa lemak tubuh Massa lemak | al per row. | OO-JO#AE1#6 | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen lemak visceral Total massa lemak tubuh Massa | al per row. | eDO-jūeAĒ1ebe | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen lemak visoeral Total massa lemak tubuh Massa lemak tubuh | al per row. | oco-joeAE1a6e | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen lemak visoeral Total massa lemak tubuh Massa lemak tubuh | al per row. | oco-joealitelo | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Total massa lemak visceral Massa lemak visceral Lingkar pinggang | al per row. | OO-JORAET so | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Class Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Total massa lemak tubuh Lingkar pinggang Lingkar | al per row. | OO-JOsAEtső | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Class Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Total massa lemak visoeral Lingkar pinggang Lingkar pinggang | al per row. | oDO-jūeAE1ethe | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Ceas Report Form |
| 7/2003, 2.43 PM<br>6. | Antropometri * Mark enly one ow BB aktual TB aktual IMT Total persen lemak tubuh Persen lemak tubuh Total massa lemak tubuh Lingkar pinggang Lingkar pinggang Rasio | al per row. | eco-joeAE1a6e | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Case Report Form |
| 7/2003, 2-43 PM<br>6. | Antropometri * Mark only one ow BB aktual TB aktual IMT Total persen lemak tubuh Total massa lemak visoeral Lingkar pinggang Lingkar pinggang | al per row. | oco-joražiteče | | 55 | | Inklusi * Check all that apply. Obese (IMT>=30 kg/m2 dan persen lemak >35%)? Etnis Sunda? Usia 18-25 thn? Tekanan darah dan gula darah puasa normal? Bersedia dan menandatangani informed | | | Case Report Form |

Kriteria



Research Ethics Committee Universitas Padjadjaran

# tificate of Attendance

NO. B03/UN6.KEP/DL/2019

This is to certify that

Prof. Dr. Ir. Hardinsyah, MS.

has attended and completed

## TRAINING ON GOOD CLINICAL PRACTICES

held in Bandung, 12 - 14 November 2019

The same of the sa

Prof. Rovina Ruslami, dr., Sp.PD., Ph.D.

Còurse Coordinator
Universitas Padjadjaran

Phamayanti, dr., Sp.A(K)., M.Kes.

of the Research Ethics Committee Universitas Padjadjaran σσασσασσασσασσασσασσασσασσασσασσασ

No: GCP-C/CRSUFMUI/06/2021/031



## CERTIFICATE OF COMPETENCE

This certificate is awarded to



### Dr. Ir. Hadi Riyadi, MS

who has passed the competency test of

### **Good Clinical Practice**

Organized by Clinical Research Supporting Unit, Faculty of Medicine, Universitas Indonesia

**Jakarta**, 10 June 2021

free

Prof. dr. Franciscus D. Suyatna, PhD, SpFK Head of CRSU FMUI